CLINICAL TRIAL: NCT01125046
Title: Phase II Trial of Bevacizumab in Patients With Recurrent or Progressive Meningiomas
Brief Title: Bevacizumab in Treating Patients With Recurrent or Progressive Meningiomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 09C2; NCI-2010-00843; STU00024715 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-05-07; First posted 2010-05-18 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-10

CONDITIONS: Acoustic Schwannoma; Adult Anaplastic Meningioma; Adult Ependymoma; Adult Grade I Meningioma; Adult Grade II Meningioma; Adult Meningeal Hemangiopericytoma; Adult Papillary Meningioma; Neurofibromatosis Type 1; Neurofibromatosis Type 2; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Neuroma, Acoustic; Meningioma; Ependymoma; Neurofibromatosis 1; Neurofibromatosis 2; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes every 2 weeks for 6 months. Patients may then receive bevacizumab IV every 3 weeks for up to 12 months. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; Avastin; recombinant humanized anti-VEGF monoclonal antibody; rhuMAb VEGF

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well bevacizumab works in treating patients with recurrent or progression meningiomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of bevacizumab in patients with recurrent or progressive benign and atypical/malignant meningiomas, despite prior therapy, as measured by six-month progression-free survival.

SECONDARY OBJECTIVES:

I. To describe the response rate and overall-survival in this patient population.

II. To evaluate the safety profile of bevacizumab in patients with recurrent meningiomas.

III. To perform an exploratory study in patients with hemangioblastoma and hemangiopericytoma.

IV. To assess tissue for VEGF and VEGFR to correlate with response. An exploratory analysis of HER-2 will be performed.

OUTLINE:

Patients receive bevacizumab IV over 30-90 minutes every 2 weeks for 6 months. Patients may then receive bevacizumab IV every 3 weeks for up to 12 months. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Criteria

* Histologically proven recurrent or progressive intracranial meningioma; this includes benign, atypical, or malignant meningioma who may or may not have neurofibromatosis type 1 or 2; pathology can be from initial surgery; OR histologically proven intracranial hemangiopericytoma, hemangioblastoma (with or without metastatic disease), acoustic neuroma, or intracranial schwannoma
* Unequivocal evidence for tumor progression by MRI (or CT scan if MRI is contraindicated); the scan must be performed within 14 days of registration
* Steroid dosing- must be on stable dose for at least 5 days prior to baseline imaging (Steroids are not required at the time of baseline imaging)
* Recent resection for recurrent tumor - patients will be eligible as long as they are greater than four weeks from surgery, have recovered from the effects of surgery, and have residual disease that can be evaluated; to best assess the extent of residual disease post-operatively, a CT/MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively; if the 96 hour scan is more than 14 days before registration, it should be repeated
* Prior radiation therapy - patients may have been treated with standard external beam radiation or radiosurgery in any combination; an interval of >= 8 weeks (56 days) must have elapsed from the completion of radiation therapy to study entry and there must be subsequent evidence of tumor progression
* Patients with prior stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based on PET, MR spectroscopy or surgical documentation of disease
* Prior therapy: there is no limitation on the number of prior surgeries, radiation therapy, radiosurgery treatments, or chemotherapy agents
* Prior surgery: must be > 4 weeks from surgery
* Prior radiation: must be 8 weeks from end of treatment
* Prior chemotherapy: must be at least 4 weeks from cytotoxic therapy and 2 weeks from biologic therapies
* All patients must sign an informed consent indicating that they are aware of the investigational nature of the study
* Patients must sign an authorization for the release of their protected health information
* Karnofsky performance status >= 60%
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 8gm/dl
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x local laboratory upper limit of normal (ULN)
* Serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x local laboratory upper limit of normal (ULN)
* Creatinine =< 2.0 mg/dl
* PT, INR, and PTT =< 1.5 times institutional upper limits of normal
* Total serum bilirubin =< 1.5
* Patients with a history of NF may have other stable CNS tumors, such as schwannoma, acoustic neuroma, or ependymoma, but ONLY if these lesions have been stable in size for the preceding 6 months
* No history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless in complete remission and off all therapy for the disease for a minimum of 5 years
* Patients may not have a history of prior treatment with inhibitors of the VEGF pathway (eg: VEGF trap, cediranib, vatalanib, sunitinib, sorafenib, etc.)
* No concurrent treatment on another clinical trial; supportive care trials or non-treatment trials, e.g. QOL, are allowed
* No history of known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
* Anticoagulation with therapeutic warfarin (INR <3) and low molecular weight heparin is allowed
* Pregnancy or breast-feeding (Patients must be surgically sterile, postmenopausal, or agree to use effective contraception during the period of therapy; the definition of effective contraception will be based on the judgment of the principal investigator or a designated associate)
* Male patients must be surgically sterile or agree to use effective contraception; women of childbearing potential must have a negative B-HCG pregnancy test documented within 14 days prior to registration
* Patient must be able to comply with the study and follow-up procedures
* Life expectancy greater than 12 weeks
* Adequately controlled hypertension (defined as systolic blood pressure =< 150 mmHg and/or diastolic blood pressure =< 100 mmHg)
* No history of hypertensive crisis or hypertensive encephalopathy
* Patients must not have New York Heart Association (NYHA) Grade II or greater congestive heart failure
* No history of myocardial infarction or unstable angina within 12 months prior to Day 1 of treatment
* No history of stroke or transient ischemic attack
* Patients must not have significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of treatment
* No history of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1 of treatment
* No evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* No history of major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of treatment or anticipation of need for major surgical procedure during the course of the study
* No history of minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1 of treatment
* No history of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1 of treatment
* Patients must not have serious non-healing wound, active ulcer, or unhealed bone fracture
* Urine protein:creatinine (UPC) ratio =< 1.0 at screening OR urine dipstick for proteinuria < 2 (patients discovered to have >= 2 proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate =< 1g of protein in 24 hours to be eligible)
* No known hypersensitivity to any component of bevacizumab
* Patients may not have a prior history of bowel perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06-17 (Actual); Primary Completion 2014-03-10 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kumthekar, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on May 19, 2010 with an accrual goal of up to 50 patients. First patient started treatment on 6/17/2010. The study was closed permanently to further enrollment on September 24, 2013 when accrual was met.
Groups:
- Treatment With Bevacizumab: Patients receive bevacizumab IV over 30-90 minutes every 2 weeks for 6 months (1 cycle = 28 days with two doses of bevacizumab). Patients may then receive bevacizumab IV every 3 weeks for up to 12 months (1 cycle = 42 days) or stay on the 2 week cycle at the discretion of the treating physician. Treatment continues in the absence of disease progression or unacceptable toxicity. After 12 months of treatment patients may continue on bevacizumab at the discretion of their treating physician.
  bevacizumab: Given IV
Period: First 6 Months of Treatment
Arm/Group | Treatment With Bevacizumab
Started | 50
Completed | 36
Not Completed | 14
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Non-compliance | 1
Not completed — Surgery | 1
Not completed — Progressive Disease | 7
Not completed — Adverse Event | 2
Period: Continued Treatment After 6 Months
Arm/Group | Treatment With Bevacizumab
Started | 36
Completed | 33
Not Completed | 3
Not completed — Progressive Disease | 2
Not completed — Adverse Event | 1
Period: Follow-up/Data Cut Off Point
Arm/Group | Treatment With Bevacizumab
Started (All patients treated on the study go into follow up period.) | 49
Completed | 16
Not Completed | 33
Not completed — Death | 29
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Bevacizumab
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
Stage of Disease (at study entry) [Count of Participants; unit: Participants] — Grading of disease was based on the degree of anaplasia, number of mitosis, and presence of necrosis using World Health Organization (WHO) classification of tumors of the central nervous system. Grades in general are as follows:
  Grade I - Benign Grade II - Atypical Grade III - Malignant
  Participants
    Stage I | 15
    Stage II | 22
    Stage III | 13
Diagnosis [Count of Participants; unit: Participants]
  Meningioma | 42
  Hemangiopericytoma | 4
  Acoustic Neuroma/Vestibular Schwannoma | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) of Patients With Recurrent or Progressive Meningiomas Treated With Bevacizumab at 6 Months
Description: Progression Free Survival (PFS) of patients with recurrent or progressive benign and atypical/malignant Meningiomas (grades I-III), despite prior therapy treated with bevacizumab will be defined from the time of registration to the study until the time of first documentation of progressive disease or death from any cause. Progressive disease will be assessed based on the Macdonald Criteria and is defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, or clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR clear worsening or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: From the start of treatment and up until 6 months of treatment or follow up
Population: PFS was analyzed based on grading of meningioma due to the difference in prognosis of grades to provide meaningful results. In general, grade I tumor grows slowly, grade II tumor grows more quickly and is often called atypical meningioma, and grade III tumor grows and spreads very quickly and is often called anaplastic or malignant meningioma.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment With Bevacizumab
Number analyzed (Participants) | 42
percentage of patients
  Grade I Meningioma: number analyzed (Participants) | 10
  Grade I Meningioma | 93 [61 to 99]
  Grade II Meningioma: number analyzed (Participants) | 21
  Grade II Meningioma | 85 [61 to 95]
  Grade III Meningioma: number analyzed (Participants) | 11
  Grade III Meningioma | 51 [22 to 75]
  Grade II/III Meningioma: number analyzed (Participants) | 32
  Grade II/III Meningioma | 73 [54 to 85]

2. Secondary Outcome: Number of Patients With Each Response
Description: Best Response of patients treated with bevacizumab with diagnosis of any of the following: meningioma, hemangiopericytoma, hemangioblastoma, acustic neuroma or schwanoma will be assessed using the MacDonald Criteria.
  In general:
  Complete Response-Complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients not on steroids.
  Partial Response-50% or greater decrease under baseline in the sum of products of perpendicular diameters of the two largest measurable lesions. No progression of evaluable disease. No new lesions.
  Stable Disease-Not CR or PR or PD. Progressive disease (PD)-25% increase in the sum of products of all measurable lesions over smallest sum observed, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR clear worsening or failure to return for evaluation due to death/deteriorating condition
Time Frame: From start of treatment and approximately every 8 weeks for up to approximately 5 years ( maximum duration any one patient was on treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Bevacizumab
Number analyzed (Participants) | 50
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 43
  Progressive Diseaase | 4
  Death | 1

3. Secondary Outcome: Safety Profile of Bevacizumab
Description: Safety of bevacizumab in patients with diagnosis of any of the following: meningioma, hemangiopericytoma, hemangioblastoma, acustic neuroma or schwanoma, will be assessed by collecting the number of adverse events experienced by patients that were determined to be at least possibly related to bevacaumab and assessed as a grade 3 or 4. AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
  In general, AEs will be graded as follows:
  Grade 1 - Mild Grade 2 - Moderate Grade 3 - Severe Grade 4 - Life-threatening Grade 5 - Fatal
Time Frame: Every 2 weeks or 3 weeks while on treatment up to 30 days after the last dose. The maximum duration any one patient was on treatment was approximately 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Bevacizumab
Number analyzed (Participants) | 50
Participants
  Hypertension | 10
  Hyponatremia | 2
  Proteinuria | 2
  Ataxia | 1
  Pancreatitis | 1
  Nausea/Vomiting | 1
  Elevated Lipase | 1
  Anemia | 1
  Infection | 1
  Muscle weakness | 1
  Epistaxis (Nosebleed) | 1
  Thrombus/embolism | 1
  Fatigue | 1

4. Secondary Outcome: Levels of VEGF, VEGRfR2 and HER2 Expression in Tumor Tissue as Compared to Response
Description: Tissue was collected for VEGF, VEGRfR2 and HER2 at baseline. Patients underwent radiological assessments every 8 weeks during treatment to determine disease status to treatment (complete response/partial response/stable disease/progressive disease). The level of VEGF, VEGRfR2 and HER2 marker expression was compared with the response as determined at the time of disease progression or death. Immunohistochemistry (IHC) will be analyzed using blobfinder technology.
  Each sample was given a score for the markers expression in the tissue 1, 2 or 3 (1=+, 2=++, 3=+++, from low to high) and a percentage 0-100% (low to high) of how much tissue it was expressed in.
  If score = 0 and percentage =0 the sample was negative for that marker. If score = 1 and percentage =10% the marker had an expression of 1 (+) in 10 percent of the tissue and so forth.
  The data is shown by patient and their best response to treatment with their score and expression for VEGF, VEGRfR2 and HER2.
Time Frame: At baseline and every 8 weeks until disease progression or death. The maximum duration any one patient was on treatment was approximately 5 years.
Measure: Number; unit: score on a scale
Arm/Group | Treatment With Bevacizumab
Number analyzed (Participants) | 42
score on a scale
  #01/Partial Response : VEGF Score | 1
  #01/Partial Response : VEGF Expression | 30
  #01/Partial Response : VEGRfR2 Score | 1
  #01/Partial Response : VEGRfR2 Expression | 10
  #01/Partial Response : HER2 Score | 0
  #01/Partial Response : HER2 Expression | 0
  #02/Stable Disease : VEGF Score | 2
  #02/Stable Disease : VEGF Expression | 80
  #02/Stable Disease : VEGRfR2 Score | 1
  #02/Stable Disease : VEGRfR2 Expression | 10
  #02/Stable Disease : HER2 Score | 1
  #02/Stable Disease : HER2 Expression | 50
  #03/Stable Disease : VEGF Score | 2
  #03/Stable Disease : VEGF Expression | 80
  #03/Stable Disease : VEGRfR2 Score | 1
  #03/Stable Disease : VEGRfR2 Expression | 20
  #03/Stable Disease : HER2 Score | 0
  #03/Stable Disease : HER2 Expression | 0
  #04/Stable Disease : VEGF Score | 2
  #04/Stable Disease : VEGF Expression | 80
  #04/Stable Disease : VEGRfR2 Score | 2
  #04/Stable Disease : VEGRfR2 Expression | 10
  #04/Stable Disease : HER2 Score | 1
  #04/Stable Disease : HER2 Expression | 10
  #07/Stable Disease : VEGF Score | 2
  #07/Stable Disease : VEGF Expression | 60
  #07/Stable Disease : VEGRfR2 Score | 2
  #07/Stable Disease : VEGRfR2 Expression | 10
  #07/Stable Disease : HER2 Score | 0
  #07/Stable Disease : HER2 Expression | 0
  #08/death : VEGF Score | 2
  #08/death : VEGF Expression | 70
  #08/death : VEGRfR2 Score | 1
  #08/death : VEGRfR2 Expression | 10
  #08/death : HER2 Score | 1
  #08/death : HER2 Expression | 30
  #09/Stable Disease : VEGF Score | 2
  #09/Stable Disease : VEGF Expression | 60
  #09/Stable Disease : VEGRfR2 Score | 0
  #09/Stable Disease : VEGRfR2 Expression | 0
  #09/Stable Disease : HER2 Score | 0
  #09/Stable Disease : HER2 Expression | 0
  #10/Stable Disease : VEGF Score | 3
  #10/Stable Disease : VEGF Expression | 70
  #10/Stable Disease : VEGRfR2 Score | 1
  #10/Stable Disease : VEGRfR2 Expression | 30
  #10/Stable Disease : HER2 Score | 0
  #10/Stable Disease : HER2 Expression | 0
  #11a/Stable Disease : VEGF Score | 3
  #11a/Stable Disease : VEGF Expression | 80
  #11a/Stable Disease : VEGRfR2 Score | 1
  #11a/Stable Disease : VEGRfR2 Expression | 10
  #11a/Stable Disease : HER2 Score | 1
  #11a/Stable Disease : HER2 Expression | 5
  #12/Stable Disease : VEGF Score | 1
  #12/Stable Disease : VEGF Expression | 20
  #12/Stable Disease : VEGRfR2 Score | 1
  #12/Stable Disease : VEGRfR2 Expression | 50
  #12/Stable Disease : HER2 Score | 0
  #12/Stable Disease : HER2 Expression | 0
  #13/Stable Disease : VEGF Score | 2
  #13/Stable Disease : VEGF Expression | 50
  #13/Stable Disease : VEGRfR2 Score | 2
  #13/Stable Disease : VEGRfR2 Expression | 70
  #13/Stable Disease : HER2 Score | 0
  #13/Stable Disease : HER2 Expression | 0
  #15/Stable Disease : VEGF Score | 2
  #15/Stable Disease : VEGF Expression | 80
  #15/Stable Disease : VEGRfR2 Score | 1
  #15/Stable Disease : VEGRfR2 Expression | 50
  #15/Stable Disease : HER2 Score | 0
  #15/Stable Disease : HER2 Expression | 0
  #16/Progressive Disease : VEGF Score | 3
  #16/Progressive Disease : VEGF Expression | 90
  #16/Progressive Disease : VEGRfR2 Score | 1
  #16/Progressive Disease : VEGRfR2 Expression | 50
  #16/Progressive Disease : HER2 Score | 0
  #16/Progressive Disease : HER2 Expression | 0
  #17/Stable Disease : VEGF Score | 3
  #17/Stable Disease : VEGF Expression | 100
  #17/Stable Disease : VEGRfR2 Score | 0
  #17/Stable Disease : VEGRfR2 Expression | 0
  #17/Stable Disease : HER2 Score | 0
  #17/Stable Disease : HER2 Expression | 0
  #19/Stable Disease : VEGF Score | 2
  #19/Stable Disease : VEGF Expression | 50
  #19/Stable Disease : VEGRfR2 Score | 1
  #19/Stable Disease : VEGRfR2 Expression | 20
  #19/Stable Disease : HER2 Score | 1
  #19/Stable Disease : HER2 Expression | 10
  #020/Stable Disease : VEGF Score | 1
  #020/Stable Disease : VEGF Expression | 80
  #020/Stable Disease : VEGRfR2 Score | 1
  #020/Stable Disease : VEGRfR2 Expression | 30
  #020/Stable Disease : HER2 Score | 1
  #020/Stable Disease : HER2 Expression | 10
  #120/Stable Disease : VEGF Score | 1
  #120/Stable Disease : VEGF Expression | 50
  #120/Stable Disease : VEGRfR2 Score | 1
  #120/Stable Disease : VEGRfR2 Expression | 10
  #120/Stable Disease : HER2 Score | 0
  #120/Stable Disease : HER2 Expression | 0
  #21/Progressive Disease : VEGF Score | 1
  #21/Progressive Disease : VEGF Expression | 70
  #21/Progressive Disease : VEGRfR2 Score | 1
  #21/Progressive Disease : VEGRfR2 Expression | 30
  #21/Progressive Disease : HER2 Score | 0
  #21/Progressive Disease : HER2 Expression | 0
  #22/Stable Disease : VEGF Score | 2
  #22/Stable Disease : VEGF Expression | 70
  #22/Stable Disease : VEGRfR2 Score | 0
  #22/Stable Disease : VEGRfR2 Expression | 0
  #22/Stable Disease : HER2 Score | 0
  #22/Stable Disease : HER2 Expression | 0
  #23/Stable Disease : VEGF Score | 2
  #23/Stable Disease : VEGF Expression | 80
  #23/Stable Disease : VEGRfR2 Score | 1
  #23/Stable Disease : VEGRfR2 Expression | 5
  #23/Stable Disease : HER2 Score | 0
  #23/Stable Disease : HER2 Expression | 0
  #26/Stable Disease : VEGF Score | 3
  #26/Stable Disease : VEGF Expression | 90
  #26/Stable Disease : VEGRfR2 Score | 2
  #26/Stable Disease : VEGRfR2 Expression | 50
  #26/Stable Disease : HER2 Score | 0
  #26/Stable Disease : HER2 Expression | 0
  #28/Stable Disease : VEGF Score | 1
  #28/Stable Disease : VEGF Expression | 50
  #28/Stable Disease : VEGRfR2 Score | 0
  #28/Stable Disease : VEGRfR2 Expression | 0
  #28/Stable Disease : HER2 Score | 0
  #28/Stable Disease : HER2 Expression | 0
  #29/Stable Disease : VEGF Score | 1
  #29/Stable Disease : VEGF Expression | 80
  #29/Stable Disease : VEGRfR2 Score | 1
  #29/Stable Disease : VEGRfR2 Expression | 20
  #29/Stable Disease : HER2 Score | 0
  #29/Stable Disease : HER2 Expression | 0
  #30/Stable Disease : VEGF Score | 2
  #30/Stable Disease : VEGF Expression | 70
  #30/Stable Disease : VEGRfR2 Score | 0
  #30/Stable Disease : VEGRfR2 Expression | 0
  #30/Stable Disease : HER2 Score | 0
  #30/Stable Disease : HER2 Expression | 0
  #31/Stable Disease : VEGF Score | 2
  #31/Stable Disease : VEGF Expression | 90
  #31/Stable Disease : VEGRfR2 Score | 0
  #31/Stable Disease : VEGRfR2 Expression | 0
  #31/Stable Disease : HER2 Score | 0
  #31/Stable Disease : HER2 Expression | 0
  #32/Stable Disease : VEGF Score | 2
  #32/Stable Disease : VEGF Expression | 80
  #32/Stable Disease : VEGRfR2 Score | 2
  #32/Stable Disease : VEGRfR2 Expression | 50
  #32/Stable Disease : HER2 Score | 1
  #32/Stable Disease : HER2 Expression | 10
  #33/Progressive Disease : VEGF Score | 3
  #33/Progressive Disease : VEGF Expression | 70
  #33/Progressive Disease : VEGRfR2 Score | 1
  #33/Progressive Disease : VEGRfR2 Expression | 10
  #33/Progressive Disease : HER2 Score | 0
  #33/Progressive Disease : HER2 Expression | 0
  #34/Stable Disease : VEGF Score | 3
  #34/Stable Disease : VEGF Expression | 70
  #34/Stable Disease : VEGRfR2 Score | 0
  #34/Stable Disease : VEGRfR2 Expression | 0
  #34/Stable Disease : HER2 Score | 0
  #34/Stable Disease : HER2 Expression | 0
  #35/Stable Disease : VEGF Score | 2
  #35/Stable Disease : VEGF Expression | 50
  #35/Stable Disease : VEGRfR2 Score | 1
  #35/Stable Disease : VEGRfR2 Expression | 50
  #35/Stable Disease : HER2 Score | 0
  #35/Stable Disease : HER2 Expression | 0
  #37/Stable Disease : VEGF Score | 3
  #37/Stable Disease : VEGF Expression | 80
  #37/Stable Disease : VEGRfR2 Score | 1
  #37/Stable Disease : VEGRfR2 Expression | 30
  #37/Stable Disease : HER2 Score | 1
  #37/Stable Disease : HER2 Expression | 5
  #38/Stable Disease : VEGF Score | 1
  #38/Stable Disease : VEGF Expression | 80
  #38/Stable Disease : VEGRfR2 Score | 1
  #38/Stable Disease : VEGRfR2 Expression | 70
  #38/Stable Disease : HER2 Score | 0
  #38/Stable Disease : HER2 Expression | 0
  #039/Stable Disease : VEGF Score | 3
  #039/Stable Disease : VEGF Expression | 100
  #039/Stable Disease : VEGRfR2 Score | 0
  #039/Stable Disease : VEGRfR2 Expression | 0
  #039/Stable Disease : HER2 Score | 0
  #039/Stable Disease : HER2 Expression | 0
  #40/Stable Disease : VEGF Score | 2
  #40/Stable Disease : VEGF Expression | 30
  #40/Stable Disease : VEGRfR2 Score | 1
  #40/Stable Disease : VEGRfR2 Expression | 50
  #40/Stable Disease : HER2 Score | 1
  #40/Stable Disease : HER2 Expression | 5
  #41/Stable Disease : VEGF Score | 2
  #41/Stable Disease : VEGF Expression | 70
  #41/Stable Disease : VEGRfR2 Score | 3
  #41/Stable Disease : VEGRfR2 Expression | 10
  #41/Stable Disease : HER2 Score | 2
  #41/Stable Disease : HER2 Expression | 10
  #42/Stable Disease : VEGF Score | 0
  #42/Stable Disease : VEGF Expression | 0
  #42/Stable Disease : VEGRfR2 Score | 0
  #42/Stable Disease : VEGRfR2 Expression | 0
  #42/Stable Disease : HER2 Score | 0
  #42/Stable Disease : HER2 Expression | 0
  #43/Stable Disease : VEGF Score | 2
  #43/Stable Disease : VEGF Expression | 50
  #43/Stable Disease : VEGRfR2 Score | 2
  #43/Stable Disease : VEGRfR2 Expression | 5
  #43/Stable Disease : HER2 Score | 0
  #43/Stable Disease : HER2 Expression | 0
  #44/Stable Disease : VEGF Score | 0
  #44/Stable Disease : VEGF Expression | 0
  #44/Stable Disease : VEGRfR2 Score | 1
  #44/Stable Disease : VEGRfR2 Expression | 10
  #44/Stable Disease : HER2 Score | 0
  #44/Stable Disease : HER2 Expression | 0
  #45/Progressive Disease : VEGF Score | 2
  #45/Progressive Disease : VEGF Expression | 30
  #45/Progressive Disease : VEGRfR2 Score | 1
  #45/Progressive Disease : VEGRfR2 Expression | 10
  #45/Progressive Disease : HER2 Score | 0
  #45/Progressive Disease : HER2 Expression | 0
  #47/Partial Response : VEGF Score | 2
  #47/Partial Response : VEGF Expression | 50
  #47/Partial Response : VEGRfR2 Score | 1
  #47/Partial Response : VEGRfR2 Expression | 50
  #47/Partial Response : HER2 Score | 0
  #47/Partial Response : HER2 Expression | 0
  #48/Stable Disease : VEGF Score | 1
  #48/Stable Disease : VEGF Expression | 50
  #48/Stable Disease : VEGRfR2 Score | 1
  #48/Stable Disease : VEGRfR2 Expression | 10
  #48/Stable Disease : HER2 Score | 0
  #48/Stable Disease : HER2 Expression | 0
  #49/Stable Disease : VEGF Score | 2
  #49/Stable Disease : VEGF Expression | 20
  #49/Stable Disease : VEGRfR2 Score | 1
  #49/Stable Disease : VEGRfR2 Expression | 70
  #49/Stable Disease : HER2 Score | 0
  #49/Stable Disease : HER2 Expression | 0
  #50/Stable Disease : VEGF Score | 2
  #50/Stable Disease : VEGF Expression | 80
  #50/Stable Disease : VEGRfR2 Score | 1
  #50/Stable Disease : VEGRfR2 Expression | 20
  #50/Stable Disease : HER2 Score | 0
  #50/Stable Disease : HER2 Expression | 0

5. Secondary Outcome: Number of Patients Alive at 1 Year, 2 Years and 3 Years Post Treatment Initiation (Overall Survival) for Patients With Recurrent or Progressive Meningiomas Treated With Bevacizumab
Description: Overall Survival (OS) of patients with Recurrent or Progressive Meningiomas Treated with Bevacizumab will be measured from the time of treatment initiation to the study until death from any cause. The raw data of number of patients documented as being alive at 1 year, 2 year, and 3 years post treatment initiation is reported here.
Time Frame: At 1 year, 2 years, 3 years post treatment initiation
Population: 2 patients were considered lost to follow up at year 2 and year 3 respectively and were not included in the numbers. Data cut off was Dec 2018 and those who had not reached 3 years are not included in the 3 year number of patients alive. No survival data was collected at these timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Bevacizumab
Number analyzed (Participants) | 50
Participants
  At 1 year | 43
  At 2 years: number analyzed (Participants) | 49
  At 2 years | 31
  At 3 years: number analyzed (Participants) | 42
  At 3 years | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of treatment initiation until 30 days post treatment discontinuation for all patients. Range of cycles of treatment completed by patients was 1-47 where one cycle equals 28 days on bevaciumab every 2 week schedule and 42 days on bevacizumab every 3 weeks. Longest time any patient was on treatment was 5 years.
Description: Data that has been collected in the database is reported here. There is still some data entry of other adverse events for a few patient being completed and this Section will be updated accordingly when all data is entered and available for reporting (if applicable).
Arm/Group | Treatment With Bevacizumab
All-Cause Mortality (participants affected / at risk) | 30/50
Serious Adverse Events (participants affected / at risk) | 22/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Bevacizumab (N=50)
Pancreatitis (Gastrointestinal disorders) | 1 — Patient with increased lipase at the time of the event
Seizure (Nervous system disorders) | 5
Anorectal Infection (Infections and infestations) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 — Patient also with ataxia and speech impairment at the time of the event
Toxic Metabolic Encephalopathy (Nervous system disorders) | 1
Epistaxis (General disorders) | 1
Aphasia (Nervous system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Left sided apraxia and numbness (Nervous system disorders) | 1
Muscle weakness and spasticity (Musculoskeletal and connective tissue disorders) | 1 — Patient also with tremors at the time of the event
Left-sided paralysis (Nervous system disorders) | 1
RPLS (Nervous system disorders) | 1
Pain: Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1
Somnolence d/t narcotic overdose (Nervous system disorders) | 1
Weakness- Lower Extremity (Musculoskeletal and connective tissue disorders) | 1
CNS Cebrovascular Ischemia (Nervous system disorders) | 1
Infection (ventriculitis) (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Viral Bronchitis (Infections and infestations) | 1
Pneymocephalus (Nervous system disorders) | 1
Wound Infection (Infections and infestations) | 1 — Patient with Pyramidal tract disturbance and gait disturbance at the time of the event
Fall (Injury, poisoning and procedural complications) | 1 — Patient had facture due to the fall
Hip Prosthesis Dislocation (Injury, poisoning and procedural complications) | 1 — Patient also with hip pain, bruising and confusion due to the event
Seizures and cognitive disturbance (Nervous system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 — Patient also with altered mental status and muscle weakness thought to be due to the event
Hemorrhage - CNS (Nervous system disorders) | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysphasia (Gastrointestinal disorders) | 1 — Patient Died during this event. Reason of death unclear
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Bevacizumab (N=50)
Anemia (Blood and lymphatic system disorders) | 3
Auditory/ear NOS (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
heaing impaired (Ear and labyrinth disorders) | 2
Blurred vision (Eye disorders) | 2
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 3
ocular vivsual other (Eye disorders) | 2
cataract (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Gastrointestinal disorders - Diarrhea (Gastrointestinal disorders) | 10
Gastrointestinal disorders - Dyspepsia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Nausea (Gastrointestinal disorders) | 16
Hemorrhage - oral cavity (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Gastrointestinal disorders - dysphagia (Gastrointestinal disorders) | 2
General disorders and administration site conditions - Edema limbs (General disorders) | 6
General disorders and administration site conditions - Fatigue (General disorders) | 21
General disorders and administration site conditions - Gait disturbance (General disorders) | 4
General disorders and administration site conditions - pain (General disorders) | 18
ear infection (Infections and infestations) | 2
Infections and infestations - other, specify (Infections and infestations) | 2
Infections and infestations -Urinary tract infection (Infections and infestations) | 3
Investigations - Alanine aminotransferase increased (Investigations) | 7
Investigations - Alkaline phosphatase increased (Investigations) | 4
Investigations - Aspartate aminotransferase increased (Investigations) | 10
Investigations - Blood bilirubin increased (Investigations) | 2
Investigations - Creatinine increased (Investigations) | 3
Investigations - Bicarbonate Serum Low (Investigations) | 2
Investigations - Lymphocyte count decreased (Investigations) | 8
Investigations - Platelet count decreased (Investigations) | 6
Neutrophil count decrease (Investigations) | 3
Investigations - Weight loss (Investigations) | 4
Investigations - White blood cell decreased (Investigations) | 8
Bruising (Injury, poisoning and procedural complications) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 19
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesmia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4
BUN elevated (Metabolism and nutrition disorders) | 2
Urine - WBCs detected (Metabolism and nutrition disorders) | 2
Urine Casts detected (Metabolism and nutrition disorders) | 3
Chloride Elevated (Metabolism and nutrition disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Teeth pain (General disorders) | 2
extremity limb pain (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness - extraocular (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness - extremity lower (Musculoskeletal and connective tissue disorders) | 3
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2
Spasicity (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Cognitive Disturbance (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 7
Dysphasia (Nervous system disorders) | 3
dysarthria (Nervous system disorders) | 7
Extrapyramidal disorder (Nervous system disorders) | 2
Headaches (Nervous system disorders) | 21
Memory impairment (Nervous system disorders) | 5
Seizure (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 5
somnolence (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 6
Agitation (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 16
renal/genitourinary - other (Renal and urinary disorders) | 2
irregular menstration (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 11
Pulmonary/ upper respiratory - otheh (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 21
Vascular other (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes